CLINICAL TRIAL: NCT03953287
Title: Pharmacokinetic/Pharmacodynamic Study of Paracetamol Taken as an Oral Chewing Capsule Versus Normal Tablet in Healthy Young Men.
Brief Title: Pharmacokinetic Study of Paracetamol.
Acronym: Para1523
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kolding Sygehus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Paracetamol1523
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Pharmacological Action
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Interventional (Clinical Trial)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacokinetic Study of Paracetamol. (Experimental): Detailed Description:
  Twelve healthy young volunteers are recruited, and the experiments begin at 07:45 after an overnight fast. BMI and blod pressure are recorded and a catheter is inserted in an antecubital vein for blood samples.
  At 08.00 participants take 500 mg paracetamol as a tablet with 200 ml tap water or a "Paracetamol1523" capsule in random order. Subsequently, blood samples are taken every minute for 3 minutes the first hour, then every 10 minutes the following two hours. In addition, blood pressure and puls rate are measured every 20 minute the first hour, and then every 30 minutes.Side effects and time to the participants registrate any effect of the drugs are assessed in a prefabricated scheme.
  The disadvantages associated with the experiment are sought monitored by adverse event registration which ends at the end of the trial. The trial day lasts 2 hours in which blood samples are taken as described above, and blood pressure and records are stored .
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — A randomized, cross over design
  Other Names: Paracetamol1523

SUMMARY:
Brief Summary:

The study evaluate the absorption rate and pharmacodynamic of different formulation of paracetamol either in the form of normal tablets or a new rapid absorbable gelation capsule formulation "Paracetamol1523" by determining T-max and area under the response curve of paracetamol in blood concentration as well as from clinical effects after intake. Data is entered on data sheet in anonymous form and processed. The results are presented in anonymous form by publication and lecture. Experts are given the supplement: "The applicant's rights in a biomedical research project

DETAILED DESCRIPTION:
Detailed Description:

Twelve healthy young volunteers are recruited, and the experiments begin at 07:45 after an overnight fast. Clinical data are recorded and a catheter is inserted in an antecubital vein for blood samples.

At 08.00 paracetamol (500 mg) taken as tablet or a "Paracetamol1523" c in random order. Subsequently, blood samples are taken every 3 minute for one hour minutes, then every 10 minutes the following two hours. In addition, blood pressure and puls rate are measured every 10 minute the first hour, and then every 30 minutes.Side effects and time to the participants registrate any effect of the drugs are assessed in a prefabricated scheme.

The disadvantages associated with the experiment are sought monitored by adverse event registration which ends at the end of the trial. The trial day lasts 4 hours in which blood samples are taken as described above, and blood pressure and records are stored .

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteers
* Must be able to swallow tablets

Exclusion Criteria:

* Diabetes
* Thyroid disease
* any medial treatment

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-08-18 (Estimated); Primary Completion 2019-12-05 (Estimated); Study Completion 2020-02-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic study of paracetamol | 4 hours
  Peak Plasma Concentration of paracetamol

SECONDARY OUTCOMES:
Pharmacokinetic study of paracetamol | 4 hours
  Area under the response curve of Paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: ole Rasmussen, M.D., Principal Investigator — Medical Dept.,Kolding Hospital, SLB, Denmark
Locations (1):
- Kolfding Sygehus, SLB, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No